CLINICAL TRIAL: NCT04439656
Title: Detecting Absence Seizures Using Eye Tracking
Status: Completed | Type: Observational
Sponsor: Rachel Kuperman (Industry)
Collaborators: Children's Hospital of Orange County (Other); University of California, San Francisco (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Rachel Kuperman, Director, Clinical Research, Eysz, Inc.
Organization: Eysz, Inc. (Industry)
Other Study IDs: DASEY
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Epilepsy, Generalized; Absence Epilepsy; Absence Seizures; Seizures; Seizure Disorder
Keywords: eye movements; seizure detection
MeSH Terms: conditions — Epilepsy, Generalized; Epilepsy, Absence; Seizures; Epilepsy | interventions — Eye-Tracking Technology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Absence Seizures: Participants with absence seizures will have their eye movements compared to the EEG recording.
  Interventions: Diagnostic Test: Eye movement analysis

INTERVENTIONS:
Diagnostic Test: Eye movement analysis — Eye movements will be analyzed to identify if seizures are present and compared to the EEG read

SUMMARY:
The goal of this study is to develop a comfortable system that uses a wearable eye-tracker similar to eyeglasses to assist people with epilepsy in counting and measuring the severity of seizures. Participants will wear an eye-tracker during a routine EEG.

DETAILED DESCRIPTION:
Seizures can be difficult to detect outside of the hospital even with careful observation by a caregiver. EEG is the best method that we have to detect seizures- but it is uncomfortable for long term use outside of the hospital. The goal of this study is to develop a comfortable system that uses a wearable eye-tracker similar to eyeglasses to assist people with epilepsy in counting and measuring the severity of seizures. People participating in this study will have a routine EEG performed while an eye tracker measures eye movements. After the EEG is complete the researchers will compare the eye movements to the EEG to develop a software program that can detect seizures from eye movements.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form- per local IRB
2. Stated willingness to comply with all study procedures including the clicker test and availability for the duration of the study
3. Male or female, aged 4-100
4. Experience known typical absence seizures as defined by the ILAE 2017 classification or referred to EEG lab for staring spell or concern for absence seizure

   a. This will allow for inclusion of children and adults across the entire spectrum of disease states including new diagnosis (medication naive), medication responsive and non-medication responsive
5. Scheduled for clinical EEG observation

Exclusion Criteria:

1. Intolerant of wearing or unable to wear the eyeglasses
2. Autism or other developmental disorder that the PI thinks will interfere with data collection
3. History of aggression that the PI thinks will interfere with data collection
4. History of not tolerating EEG that the PI thinks will interfere with data collection
5. Unable to give consent (for individuals ≥ 18 years old) unless they have an adult with power of attorney to consent

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children or adults with absence seizures.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Eysz algorithm to detect absence seizures | 1 hour
  EEG is burdensome and limited. The current accepted method of counting seizures is observation which fails to identify > 50% of seizures. The goal is to validate the Eysz absence seizure detection algorithm and show significant improvement over current standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kuperman, MD, Principal Investigator — Eysz, Inc.
Locations (5):
- United States (5):
  - Children's Hospital Orange County, Orange, California
  - Rady Children's Hospital, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Texas Child Neurology, Plano, Texas

IPD SHARING:
Plan to Share IPD: No